CLINICAL TRIAL: NCT01900483
Title: Brain Functions in Patients Before and After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Sabine Frank, Dr., University Hospital Tuebingen
Other Study IDs: BSD
Record Dates: First submitted 2013-07-08; First posted 2013-07-16 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- pre bariatric surgery
- post bariatric surgery

SUMMARY:
The project will specifically focus on the examination of the influence of substantial weight loss due to bariatric surgery on brain functions. Our hypothesis is that substantial weight loss after Bariatric Surgery (BS) is also accompanied by changes in the balance of reward and inhibitory networks in diabetic subjects. Therefore the investigators will conduct a functional magnetic resonance imaging (fMRI) study investigating functional measures.

ELIGIBILITY:
Inclusion Criteria:

* bariatric surgery in the past or in the future
* diabetes (at least before surgery)

Exclusion Criteria:

* fMRI contraindications
* claustrophobia

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: volunteers pre and post bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Differential brain functions | at least 6 months after bariatric surgery (experimental group)
  brain functions will be measured by blood oxygen level dependent effects

OTHER OUTCOMES:
Behavioral measurements | pre surgery (group 1) and at least 6 months after surgery
  eating behavior

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Tuebingen, MEG Center, Tübingen, Germany

REFERENCES:
- [Derived] Frank S, Heinze JM, Fritsche A, Linder K, von Feilitzsch M, Konigsrainer A, Haring HU, Veit R, Preissl H. Neuronal Food Reward Activity in Patients With Type 2 Diabetes With Improved Glycemic Control After Bariatric Surgery. Diabetes Care. 2016 Aug;39(8):1311-7. doi: 10.2337/dc16-0094. Epub 2016 Jun 12. PMID 27293200